CLINICAL TRIAL: NCT01630837
Title: Frequency of Oral Hygiene in the Maintenance of Gingival Health
Brief Title: Frequency of Oral Hygiene
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Santa Maria (Other)
Responsible Party: Principal Investigator, Tatiana Militz Perrone Pinto, Frequency of oral hygiene in the maintenace of gingival health, Universidade Federal de Santa Maria
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: FHB0186.0.243.000-10
Record Dates: First submitted 2012-06-26; First posted 2012-06-28 (Estimated); Last update posted 2012-06-28 (Estimated); Status verified 2012-06

CONDITIONS: Gingivitis; Oral Health
MeSH Terms: conditions — Gingivitis

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 12h (Other): Frequency of oral hygiene was 12 to 12 hours.
  Interventions: Other: frequency of oral hygiene
- 24h (Other): Frequency of oral hygiene was 24 to 24 hours.
  Interventions: Other: frequency of oral hygiene
- 48h (Other): Frequency of oral hygiene was 48 to 48 hours.
  Interventions: Other: frequency of oral hygiene
- 72h (Other): Frequency of oral hygiene was 72 to 72 hours.
  Interventions: Other: frequency of oral hygiene

INTERVENTIONS:
Other: frequency of oral hygiene — the frequency of oral hygiene was 12 to 12 hours, 24 to 24 hours, 48 to 48 hours and 72 to 72 hours.

SUMMARY:
The purpose of this study is to evaluate the frequency of oral hygiene in the maintenance of gingival health in patients with an adequate method of oral hygiene.

DETAILED DESCRIPTION:
The study was a randomized blinded clinical trial. Eligible patients underwent a pre-clinical period in order to eliminate factors that could interfere with the proper plaque control. Forty-five non dental students with healthy gingival (maximum 5% of sites showing gingival bleeding) were randomized into four groups according to the frequency of oral hygiene (every 12h, 24h, 48h or 72h). Plaque Index (PLI) and Gingival Index (GI) were evaluated by two trained examiners at baseline, 15 days and 30 days.

ELIGIBILITY:
Inclusion Criteria:

* students of graduate courses at the Federal University of Santa Maria and Franciscan University Center
* a minimum age of 18 years
* filling all space interdental papilla
* at least 24 teeth
* maximum 15% of sites with gingivitis.

Exclusion Criteria:

* dental students
* pregnant woman
* diabetics
* smokers
* orthodontic equipment
* antimicrobial prophylaxis
* antibiotic
* anti-inflammatory
* psychomotor disturbances
* periodontitis
* PD ≥ 3mm

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2011-05; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
gingivitis expressed as an increase in mean gingival index in the experimental period | one month of evaluetion

SECONDARY OUTCOMES:
changes in plaque levels and variations of the average percentage of sites with different GI scores during the study | one month of evaluetion

CONTACTS AND LOCATIONS:
Locations (1):
- Federal University of Santa Maria, Santa Maria, Rio Grande do Sul, Brazil

REFERENCES:
- [Derived] de Freitas GC, Pinto TM, Grellmann AP, Dutra DA, Susin C, Kantorski KZ, Moreira CH. Effect of self-performed mechanical plaque control frequency on gingival inflammation revisited: a randomized clinical trial. J Clin Periodontol. 2016 Apr;43(4):354-8. doi: 10.1111/jcpe.12520. Epub 2016 Mar 29. PMID 26823235
- [Derived] Pinto TM, de Freitas GC, Dutra DA, Kantorski KZ, Moreira CH. Frequency of mechanical removal of plaque as it relates to gingival inflammation: a randomized clinical trial. J Clin Periodontol. 2013 Oct;40(10):948-54. doi: 10.1111/jcpe.12135. Epub 2013 Aug 2. PMID 23909568